CLINICAL TRIAL: NCT06286423
Title: Colchicine in Acutely Decompensated Heart Failure With Reduced Ejection Fraction: a Pilot Study
Brief Title: Colchicine in Acutely Decompensated HFREF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Antonio Abbate, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSR220446
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure; Decompensated Heart Failure; Heart Failure With Reduced Ejection Fraction
Keywords: Colchicine; Heart Failure; Decompensated Heart Failure; Heart Failure with Reduced Ejection Fraction; HFrEF
MeSH Terms: conditions — Heart Failure | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: The study team is planning to use controls in the present study. Controls will be patients from the target population, i.e. acutely decompensated heart failure with reduced ejection fraction.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine 0.6 mg treatment group (Experimental): Treatment group will be given active drug (0.6mg Colchicine) 2x/day (once if subject has kidney disease) for 14 days. Subsequently treatment group subjects will be given active drug (0.6mg Colchicine) 1x/day for 76 +/- days (or once every other day if subject has kidney disease).
  Interventions: Drug: Colchicine 0.6 mg
- Control/Placebo group (Placebo Comparator): Control/Placebo group will be given placebo that looks identical to study drug with no active ingredients and will take 2x/day (once if subject has kidney disease) for 14 days. Subsequently Control/Placebo group will be given placebo 1x/day for 76 +/- days (or once every other day if subject has kidney disease).
  Interventions: Drug: Control/Placebo group

INTERVENTIONS:
Drug: Colchicine 0.6 mg — Colchicine treated subjects will take 0.6mg of drug 2x per day (1 time if kidney disease is present) for 14 days, then will take 0.6mg of drug 1x per day (or every other day if kidney disease is present) for 76 +/1 days.
  Other Names: Colcrys; Gloperba; Lodoco; Mitigare
  Arms: Colchicine 0.6 mg treatment group
Drug: Control/Placebo group — Placebo treated subjects will take 0.6mg of placebo 2x per day (1 time if kidney disease is present) for 14 days, then will take 0.6mg of placebo1x per day (or every other day if kidney disease is present) for 76 +/1 days.
  Arms: Control/Placebo group

SUMMARY:
This is a double blind, placebo-controlled pilot trial randomizing patients admitted to the hospital with acutely decompensated heart failure (ADHF) and inflammation to receive either colchicine or matching placebo.

Upon enrollment, patients will be randomized 1:1 to receive either the experimental drug (Colchicine) or matching placebo. The regimen in the active arm will consist of 14 days of Colchicine 0.6 mg bid followed by 76±14 days of Colchicine 0.6 mg once per day. Placebo regimen will be analogous, with one pill bid for 14 days followed by one pill once per day for 76 days. Dose reduction for patients with Stage III chronic kidney disease is allowed as detailed in the protocol. At the same time, dose reduction can also be elected in case of GI symptoms. The study team will transiently stop the experimental medication in case of acute kidney injury (AKI), defined per Kidney Disease Improving Global Outcomes (KDIGO) Stage I, as specified in the protocol.

These patients will continue with their standard of care for the management of heart failure which consists of a combination of medications that relieve congestion, normalize blood pressure and heart rate, and block the effects of hormones on the heart. The proposed treatment will be in addition to standard of care. No standard of care medications will be withheld. While inflammation is a known risk factor in heart failure, there are no standard anti-inflammatory drugs used in patients with heart failure, as the benefit is not established. The study team will study colchicine, an anti-inflammatory drug, as compares with placebo.

Blood will be obtained from the patients in order to measure hsCRP and IL-6. Blood samples will be collected at baseline, 24±6h, 48±6h and 72±6h after treatment initiation, and subsequently at 14±7 days and at study closure. The first four blood samples will be obtained while the subject is still admitted to the hospital. The blood sample at 14±7 days will be obtained during an outpatient encounter. A study closure visit with clinical assessment and experimental drug collection for capsule counting to assess compliance will be conducted at 90±14; the final blood sample will be collected at that time.

DETAILED DESCRIPTION:
Colchicine - a pleotropic anti-inflammatory drug Colchicine is a natural alcaloid extract from plants of the genus Colchium (autumn crocus). From a pharmacological point of view, colchicine binds in a poorly reversible manner to tubulin and prevents microtubule formation, therefore interfering with organelle trafficking, intercellular adhesion and cellular migration. Interestingly, colchicine at therapeutic concentration was shown to inhibit nucleotide-binding oligomerization domain, leucine-rich repeat-containing protein (NLRP) 3 inflammasome, hence inhibit the release of interleukin-1 (IL-1), to reduce the surface expression and downstream signaling of tumor necrosis factor (TNF) and alter leukocyte and endothelial expression of L-selectin and E-selecting respectively, potentially interfering with leukocytes homing and extravasation. The net effect is a potently anti-inflammatory, which lead to successful use of colchicine in the treatment of primarily inflammatory condition, in particular acute arthritis such as gout or pseudogout, and serositis.

Colchicine in cardiovascular disease The positive effects of colchicine in cardiovascular conditions have long been appreciated. In particular, colchicine has been successfully used to resolve pericardial inflammation, and eventually symptoms, in pericarditis, and to effectively prevent recurrences in those individuals who develop recurrent pericarditis. More recent data have shown a significant reduction of recurrent myocardial infarction (MI) and stroke with low dose colchicine among patient with recent MI, possibly due to resolution of "vulnerable" plaque phenotype or prevention of plaque activation in the setting of an acute inflammatory condition. Interestingly, a recent meta-analysis showed that low dose colchicine was in fact able to significantly abate systemic inflammation among patients with chronic coronary artery disease. Of note, the effect was most pronounced among patients with baseline high-sensitivity C-reactive protein (hs-CRP) ≥3.0 mg/l and for treatment duration over 7 days, and was higher for doses of 1.0 mg daily than lower colchicine doses.

Heart failure is an inflammatory condition Inflammation promotes and aggravates heart failure (HF). Of note, master inflammatory cytokines, in particular interleukin-1 (IL-1) was shown to cause direct cardio-depression and induce myocyte contractile dysfunction in both humans and pre-clinical models of cardiovascular diseases. Of note, elevated levels of inflammation and sustained subclinical inflammation over time is associated with worse HF outcomes. After a HF exacerbation, patients are at higher risk of further decompensation. Such time window lasts approximately 30 to 90 days and has been defined the vulnerable period of HF. Given that elevated inflammatory burden has been associated with early HF adverse events, it is possible, although yet unproven, that inflammation could play a role in the vulnerable period.

Targeted inhibition of inflammatory pathways was shown to abate systemic inflammation in HF patients, and to improve cardiovascular performance in terms of exercise capacity and peak VO2 on cardiopulmonary exercise tests. A single-center randomized controlled trial randomizing 267 patients with HF with reduced ejection fraction, who were clinically stable, to receive either placebo or colchicine showed a significant reduction of inflammatory biomarkers, namely high sensitivity C-reactive protein (hsCRP) and interleukin 6 (IL-6). No reduction in mortality or HF-related hospitalization was observed, but a trend towards improved subjective symptoms was observed. Of note, the study did not include patients with recently decompensated HF, which are the ones who show signs of greater systemic inflammation, are at increased risk for adverse outcomes and are most likely to significantly benefit from additional treatments. In the prior study, patients were indeed not selected according to baseline levels of inflammation. In particular, epidemiological studies have shown how higher baseline levels of inflammation are associated with worse HF prognosis, and our group has shown that HFrEF patients with high inflammatory burden at baseline are likely to benefit from modulation of inflammation. More recently, a retrospective, single-center study performed at University of Virginia showed that among 1047 patients admitted for acutely decompensated HF (ADHF) those (N=237) who were chronically on Colchicine for other, non-cardiac reasons, i.e. crystal arthropathy, had significantly better in-hospital outcomes when compared to HF patient who did not chronically receive colchicine (N=810). Of note, this appears to be the largest study to assess the effects of colchicine in this population and suggesting a promising therapeutic role for colchicine in ADHF.

Because elevated levels of clinical and subclinical inflammation are associated with worse outcomes and since patients are at higher risk of further decompensation within 30 to 90 days after an episode of HF, a 90 day dosing window was chosen. Unfortunately, no data on the effect of colchicine on the vulnerable period (first 90 days after the acute episode) was available in the prior study.

The investigators hypothesize that treatment with colchicine is safe to start in patients with acutely decompensated HF, and it will significantly inhibit systemic inflammation, as shown by a reduction of biomarkers of systemic inflammation, i.e. hsCRP, in patients with acutely decompensated HF with reduced left ventricular ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

1. Primary admission diagnosis of acute decompensated heart failure as evidenced by:

   * Heart failure symptoms and at least one of the following:
   * Pulmonary congestion/edema at physical exam (or chest radiography)
   * E/e' > 13 on transthoracic echocardiography
   * Left heart catheterization showing elevated left ventricular (LV) end-diastolic pressure >18 mmHg or right heart catheterization showing pulmonary artery occluding pressure (wedge) >16 mmHg
   * Elevated plasma B-type natriuretic peptide (>100 pg/ml) or N-terminal B-type natriuretic peptide (>300 pg/ml)
2. LV systolic dysfunction (left ventricular ejection fraction [LVEF] <40%) during the index hospitalization or prior 12 months;
3. Expected duration of heart failure at least three months
4. Age 18 years or older
5. Willing and able to provide written informed consent
6. Screening plasma CRP >0.3 mg/dL (3 mg/L) or high-sensitivity CRP >2 mg/L

Exclusion Criteria:

1. Concomitant clinically significant comorbidities that would interfere with the execution or interpretation of the study, including but not limited to acute coronary syndromes, uncontrolled hypertension or orthostatic hypotension, tachy- or brady-arrhythmias, acute or chronic pulmonary disease or neuromuscular disorders affecting respiration
2. Cardiac resynchronization therapy (CRT), coronary artery revascularization procedures, or heart valve surgeries performed within 3 months or planned during the admission
3. Previous or planned implantation of left ventricular assist devices or heart transplantation
4. Chronic use of intravenous inotropes
5. Current or recent (i.e. within 4 half-lives) use of immunosuppressive or anti-inflammatory drugs (not including NSAIDs).
6. Current treatment with colchicine or planned initiation of colchicine therapy in the next three months for gout
7. Chronic inflammatory disorder, including but not limited to rheumatoid arthritis and systemic lupus erythematosus
8. Active infection (of any type)
9. Chronic or recurrent infectious disease, including hepatitis B virus, hepatitis C virus, and HIV/AIDS
10. Prior (within the past 5 years) or current malignancy, with the exclusion of in situ lesion with low potential for progression
11. Any comorbidity leading to expected survival less than three months or inability to complete the study
12. End-stage kidney disease requiring renal replacement therapy
13. Neutropenia (<2,000/mm3) or Thrombocytopenia (<50,000/mm3)
14. Pregnancy

    * For all biological females with child bearing potential a pregnancy test will be performed as part of standard of care.
15. Presence of specific contraindications to colchicine treatment, which may include

    * Previous adverse reaction to colchicine
    * Biliary obstruction
    * Renal impairment with estimated glomerular filtration rate (eGFR) <30 ml/min
    * Liver cirrhosis from stage Child-Pugh A to more advanced
16. Prisoners
17. Treatment with medication contraindicated for concomitant use with colchicine per

Food and Drugs Administration labeling, including:

* Protease inhibitors
* Macrolides antibiotic
* Ketoconazole, Fluconazole and Itraconazole
* Nefazodone
* Non-dihydropiridine calcium channel blockers
* Aprepitant
* Ranolazine
* Cyclosporine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Difference in the change in high sensitivity C-reactive protein (hsCRP) between colchicine arm and placebo arm in the first 72 hours of treatment | Baseline to 72 hours
  Change in plasma concentration of hsCRP between baseline and after 72 hours after treatment initiation, comparing colchicine arm vs placebo

SECONDARY OUTCOMES:
Difference in hsCRP area under curve between colchicine and placebo arm at 14 days | Baseline to 14 days
  Area under curve of hsCRP measurements obtained at baseline, 24h, 48h, 72h and 14 days, comparing colchicine vs placebo
Difference in change in plasma IL-6 concentration between colchicine arm and placebo arm in the first 72 hours of treatment | Baseline to 72 hours
  Change in plasma concentration of IL-6 between baseline and after 72 hours after treatment initiation, comparing colchicine arm vs placebo

OTHER OUTCOMES:
Difference in the incidence of a composite of all-cause mortality or hospitalizations for heart failure at 90 days | Baseline to 90 days
  Occurrence of death or heart failure hospitalization during trial participation, comparing colchicine and placebo arms

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Abbate, MD, Principal Investigator — UVA Health
Locations (1):
- UVA Health, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Dalbeth N, Lauterio TJ, Wolfe HR. Mechanism of action of colchicine in the treatment of gout. Clin Ther. 2014 Oct 1;36(10):1465-79. doi: 10.1016/j.clinthera.2014.07.017. Epub 2014 Aug 21. PMID 25151572
- [Background] Leung YY, Yao Hui LL, Kraus VB. Colchicine--Update on mechanisms of action and therapeutic uses. Semin Arthritis Rheum. 2015 Dec;45(3):341-50. doi: 10.1016/j.semarthrit.2015.06.013. Epub 2015 Jun 26. PMID 26228647
- [Background] Pascart T, Richette P. Colchicine in Gout: An Update. Curr Pharm Des. 2018;24(6):684-689. doi: 10.2174/1381612824999180115103951. PMID 29336252
- [Background] Aviel YB, Rawan S, Fahoum S, Wexler I, Berkun Y. Discontinuation of Colchicine Therapy in Children With Familial Mediterranean Fever. J Rheumatol. 2021 Nov;48(11):1732-1735. doi: 10.3899/jrheum.201158. Epub 2021 May 15. PMID 33993110
- [Background] Bayes-Genis A, Adler Y, de Luna AB, Imazio M. Colchicine in Pericarditis. Eur Heart J. 2017 Jun 7;38(22):1706-1709. doi: 10.1093/eurheartj/ehx246. No abstract available. PMID 30052886
- [Background] Imazio M, Brucato A, Cemin R, Ferrua S, Maggiolini S, Beqaraj F, Demarie D, Forno D, Ferro S, Maestroni S, Belli R, Trinchero R, Spodick DH, Adler Y; ICAP Investigators. A randomized trial of colchicine for acute pericarditis. N Engl J Med. 2013 Oct 17;369(16):1522-8. doi: 10.1056/NEJMoa1208536. Epub 2013 Aug 31. PMID 23992557
- [Background] Tardif JC, Kouz S, Waters DD, Bertrand OF, Diaz R, Maggioni AP, Pinto FJ, Ibrahim R, Gamra H, Kiwan GS, Berry C, Lopez-Sendon J, Ostadal P, Koenig W, Angoulvant D, Gregoire JC, Lavoie MA, Dube MP, Rhainds D, Provencher M, Blondeau L, Orfanos A, L'Allier PL, Guertin MC, Roubille F. Efficacy and Safety of Low-Dose Colchicine after Myocardial Infarction. N Engl J Med. 2019 Dec 26;381(26):2497-2505. doi: 10.1056/NEJMoa1912388. Epub 2019 Nov 16. PMID 31733140
- [Background] Pan Z, Cheng J, Yang W, Chen L, Wang J. Effect of colchicine on inflammatory markers in patients with coronary artery disease: A meta-analysis of clinical trials. Eur J Pharmacol. 2022 Jul 15;927:175068. doi: 10.1016/j.ejphar.2022.175068. Epub 2022 May 27. PMID 35644423
- [Background] Van Tassell BW, Toldo S, Mezzaroma E, Abbate A. Targeting interleukin-1 in heart disease. Circulation. 2013 Oct 22;128(17):1910-23. doi: 10.1161/CIRCULATIONAHA.113.003199. No abstract available. PMID 24146121
- [Background] Abbate A, Toldo S, Marchetti C, Kron J, Van Tassell BW, Dinarello CA. Interleukin-1 and the Inflammasome as Therapeutic Targets in Cardiovascular Disease. Circ Res. 2020 Apr 24;126(9):1260-1280. doi: 10.1161/CIRCRESAHA.120.315937. Epub 2020 Apr 23. PMID 32324502
- [Background] Golino M, Moroni F, Abbate A. Connecting the Dots: Inflammatory Burden and Outcomes in Heart Failure. J Am Heart Assoc. 2023 Oct 3;12(19):e031786. doi: 10.1161/JAHA.123.031786. Epub 2023 Sep 30. No abstract available. PMID 37776202
- [Background] Gracia E, Singh P, Collins S, Chioncel O, Pang P, Butler J. The Vulnerable Phase of Heart Failure. Am J Ther. 2018 Jul/Aug;25(4):e456-e464. doi: 10.1097/MJT.0000000000000794. No abstract available. PMID 29985824
- [Background] Alonso-Martinez JL, Llorente-Diez B, Echegaray-Agara M, Olaz-Preciado F, Urbieta-Echezarreta M, Gonzalez-Arencibia C. C-reactive protein as a predictor of improvement and readmission in heart failure. Eur J Heart Fail. 2002 Jun;4(3):331-6. doi: 10.1016/s1388-9842(02)00021-1. PMID 12034159
- [Background] Van Tassell BW, Trankle CR, Canada JM, Carbone S, Buckley L, Kadariya D, Del Buono MG, Billingsley H, Wohlford G, Viscusi M, Oddi-Erdle C, Abouzaki NA, Dixon D, Biondi-Zoccai G, Arena R, Abbate A. IL-1 Blockade in Patients With Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2018 Aug;11(8):e005036. doi: 10.1161/CIRCHEARTFAILURE.118.005036. PMID 30354558
- [Background] Trankle CR, Canada JM, Cei L, Abouzaki N, Oddi-Erdle C, Kadariya D, Christopher S, Viscusi M, Del Buono M, Kontos MC, Arena R, Van Tassell B, Abbate A. Usefulness of Canakinumab to Improve Exercise Capacity in Patients With Long-Term Systolic Heart Failure and Elevated C-Reactive Protein. Am J Cardiol. 2018 Oct 15;122(8):1366-1370. doi: 10.1016/j.amjcard.2018.07.002. Epub 2018 Jul 20. PMID 30244844
- [Background] Deftereos S, Giannopoulos G, Panagopoulou V, Bouras G, Raisakis K, Kossyvakis C, Karageorgiou S, Papadimitriou C, Vastaki M, Kaoukis A, Angelidis C, Pagoni S, Pyrgakis V, Alexopoulos D, Manolis AS, Stefanadis C, Cleman MW. Anti-inflammatory treatment with colchicine in stable chronic heart failure: a prospective, randomized study. JACC Heart Fail. 2014 Apr;2(2):131-7. doi: 10.1016/j.jchf.2013.11.006. PMID 24720919
- [Background] Van Tassell BW, Raleigh JM, Abbate A. Targeting interleukin-1 in heart failure and inflammatory heart disease. Curr Heart Fail Rep. 2015 Feb;12(1):33-41. doi: 10.1007/s11897-014-0231-7. PMID 25315037
- [Background] Van Tassell BW, Canada J, Carbone S, Trankle C, Buckley L, Oddi Erdle C, Abouzaki NA, Dixon D, Kadariya D, Christopher S, Schatz A, Regan J, Viscusi M, Del Buono M, Melchior R, Mankad P, Lu J, Sculthorpe R, Biondi-Zoccai G, Lesnefsky E, Arena R, Abbate A. Interleukin-1 Blockade in Recently Decompensated Systolic Heart Failure: Results From REDHART (Recently Decompensated Heart Failure Anakinra Response Trial). Circ Heart Fail. 2017 Nov;10(11):e004373. doi: 10.1161/CIRCHEARTFAILURE.117.004373. PMID 29141858
- [Background] Roth ME, Chinn ME, Dunn SP, Bilchick KC, Mazimba S. Association of colchicine use for acute gout with clinical outcomes in acute decompensated heart failure. Clin Cardiol. 2022 Jul;45(7):733-741. doi: 10.1002/clc.23830. Epub 2022 Apr 28. PMID 35481608
- [Background] Van Tassell BW, Abouzaki NA, Oddi Erdle C, Carbone S, Trankle CR, Melchior RD, Turlington JS, Thurber CJ, Christopher S, Dixon DL, Fronk DT, Thomas CS, Rose SW, Buckley LF, Dinarello CA, Biondi-Zoccai G, Abbate A. Interleukin-1 Blockade in Acute Decompensated Heart Failure: A Randomized, Double-Blinded, Placebo-Controlled Pilot Study. J Cardiovasc Pharmacol. 2016 Jun;67(6):544-51. doi: 10.1097/FJC.0000000000000378. PMID 26906034
- [Background] Kajikawa M, Higashi Y, Tomiyama H, Maruhashi T, Kurisu S, Kihara Y, Mutoh A, Ueda SI. Effect of short-term colchicine treatment on endothelial function in patients with coronary artery disease. Int J Cardiol. 2019 Apr 15;281:35-39. doi: 10.1016/j.ijcard.2019.01.054. Epub 2019 Jan 15. PMID 30683457

DOCUMENTS (1):
  • Informed Consent Form (2024-01-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT06286423/ICF_000.pdf